CLINICAL TRIAL: NCT00318266
Title: NMP22 Provides Improved Sensitivity in Detecting Bladder Cancers
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: R-05-885; 11720E
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2008-11

CONDITIONS: Bladder Cancer
Keywords: Detection of Bladder Cancer using NMP22 Urine Test Kit
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with suerficial transitional cell carcinoma
  Interventions: Device: Nuclear Matrix Protein 22 Urine sample kit

INTERVENTIONS:
Device: Nuclear Matrix Protein 22 Urine sample kit — Urine sample obtained from patient will be tested with the NMP22 sample kit to see if it can detect bladder cancer.

SUMMARY:
It is hypothesized that the NMP22(Nuclear Matrix Protein) Bladder Check ® Test will demonstrate improved sensitivity over that of standard urine cytology for patients with superficial transitional cell carcinoma at high risk of recurrence.

DETAILED DESCRIPTION:
Patients who have been previously treated for bladder cancer and are at a high risk for recurrence are being monitored for recurrence every 3 months with urine cytology and cystoscopy as part of standard care.The NMP22 Bladder Cancer ® Test Kit has been designed to provide an alternative to regular urine cytology. A urine sample will be provided and divided with a portion being used to assess the NMP22 test kit and the remaining sample to be sent to the lab for regular urine cytology. Patient charts will be reviewed by a medical student to record age, clinical stage, pathologic stage, time to disease progression/recurrence, site of recurrence and survival data.

ELIGIBILITY:
Inclusion Criteria:

* · History of pTis, pT1, large (>2cm) pTa or multiple pTa bladder cancer tumours.

Written Informed Consent prior to any study-related procedures.

Exclusion Criteria:

* History of bladder cancer tumours other than those listed in inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a history og pTis, pT1, larger ( >2 cm) pTa or multiple pTa bladder tumors.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Izawa, MD FRCSC, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada